CLINICAL TRIAL: NCT00019240
Title: PHASE II PROTOCOL WITH LABORATORY CORRELATES OF 1-[(S)-3-HYDROXY-2-(PHOSPHOMETHOXY)PROPYL]CYTOSINE DIHYDRATE(CIDOFOVIR) IN PATIENTS WITH KAPOSI'S SARCOMA (KS)
Brief Title: Antiviral Therapy in Treating Patients With Kaposi's Sarcoma With or Without HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065260; NCI-97-C-0024C; NCT00001559 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2004-04-21 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2007-11

CONDITIONS: Sarcoma
Keywords: classic Kaposi sarcoma; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Cidofovir

INTERVENTIONS:
Drug: cidofovir

SUMMARY:
RATIONALE: Herpesvirus is found in Kaposi's sarcoma lesions in most patients; it is therefore possible that the herpesvirus has a role in causing Kaposi's sarcoma. Cidofovir is an antiviral drug that acts against many types of herpesvirus, and may be an effective treatment for Kaposi's sarcoma.

PURPOSE: Phase II trial to study the effectiveness of cidofovir in treating patients with Kaposi's sarcoma with or without HIV infection.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of intravenous cidofovir in patients with Kaposi's sarcoma (KS) with and without human immunodeficiency virus (HIV) infection. II. Assess the effect of intravenous cidofovir on the load of KS-associated herpesvirus/human herpesvirus-8 in KS lesions and peripheral blood mononuclear cells by quantitative polymerase chain reaction. III. Assess the toxicity of cidofovir in KS patients with and without HIV infection. IV. Assess the effect of cidofovir on angiogenic cytokines related to the pathogenesis of KS.

OUTLINE: All patients receive intravenous cidofovir weekly for 2 weeks, then every other week for 6 months. Patients with a complete or partial response may continue treatment until disease progression intervenes.

PROJECTED ACCRUAL: Up to 25 evaluable patients will be entered over approximately 6 months if there are at least 2 responses in the first 15 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven Kaposi's sarcoma (KS) HIV infection (measured by ELISA and Western blot) allowed NCI pathology review required At least 5 measurable lesions required No prior local therapy to indicator lesions Lesions evaluable by noninvasive methods No actively bleeding or critically located KS of immediate risk to patient or at the discretion of the Principal Investigator and/or Study Chairperson No pulmonary or other potentially acutely life-threatening KS lesions

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: More than 3 months Hematopoietic: Absolute neutrophil count at least 750/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 11 g/dL (10 g/dL in women) CD4 count greater than 50 cells per cubic millimeter Hepatic: Bilirubin no greater than 1.5 times normal (unless due to Gilbert's disease) Patients on protease inhibitors may have bilirubin no greater than 3.5 mg/dL (direct bilirubin no greater than 0.2 mg/dL) AST/ALT no greater than 75 IU/mL Alkaline phosphatase no greater than 2.5 times normal Renal: Creatinine less than 1.5 mg/dL Creatinine clearance (calculated) greater than 55 mL/min Proteinuria less than 2+ Cardiovascular: No significant EKG abnormality Other: No actively life-threatening infection At least 14 days since treatment for serious infection No known clinically significant allergy to probenecid or sulfa No grade 3 or worse clinical or laboratory toxicity other than lymphopenia No medical condition that precludes protocol treatment or informed consent No second malignancy within 1 year except basal cell skin cancer No pregnant or nursing women Negative pregnancy test required of fertile women within 1 week prior to entry, every 4 weeks while on study, and 4 weeks after last treatment Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: At least 1 week since treatment with any of the following: Diuretics Vidarabine Amphotericin B Aminoglycoside antibiotics Intravenous pentamidine Other known or potentially nephrotoxic agents Other investigational agents with anti-herpesvirus activity At least 4 weeks since systemic or local anti-herpesvirus therapy other than mucocutaneous acyclovir cream At least 4 weeks since systemic therapy for KS or other systemic or cutaneous malignancy At least 1 month since discontinuation of antiretroviral therapy Concurrent antiretroviral therapy allowed provided doses of the following, either alone or in combination, stable for at least 1 month prior to entry: AZT ddC 3TC ddI d4T protease inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-11; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kedes DH, Ganem D. Sensitivity of Kaposi's sarcoma-associated herpesvirus replication to antiviral drugs. Implications for potential therapy. J Clin Invest. 1997 May 1;99(9):2082-6. doi: 10.1172/JCI119380. PMID 9151779